CLINICAL TRIAL: NCT00440869
Title: Effects of N-acetylcysteine on Muscle Fatigue in ESRD
Brief Title: Effects of N-acetylcysteine on Muscle Fatigue in Hemodialysis
Acronym: NAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Kirsten Johansen, MD, NCIRE, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21-DK077350 (completed); DK-077350-01; R21DK077350 (NIH)
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-03

CONDITIONS: End-Stage Renal Disease; Dialysis; Hemodialysis
Keywords: N-acetylcysteine; oxidative stress; muscle fatigue; end-stage renal disease; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-acetylcysteine (Experimental): Active
  Interventions: Dietary Supplement: N-acetylcysteine
- placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: N-acetylcysteine — 600 mg po bid
  Arms: N-acetylcysteine
Dietary Supplement: placebo — bid oral dosing
  Arms: placebo

SUMMARY:
The purposes of the study are to determine whether oxidative stress causes the muscle of dialysis patients to tire more quickly than muscle of people without kidney disease and to determine whether treatment with N-acetylcysteine, an antioxidant, can improve muscle endurance.

DETAILED DESCRIPTION:
Muscle dysfunction is a major problem for patients with end-stage renal disease (ESRD). Specifically, these patients experience approximately three-fold greater muscle fatigue of the lower extremities during intermittent submaximal contractions than healthy control subjects. Thus, a treatment that could ameliorate muscle fatigue in this population has the potential to increase endurance during activities of daily living and improve quality of life. Dialysis patients have been shown to have high levels of various markers of oxidative stress, and oxidative stress has been associated with excessive muscle fatigue in other patient populations, but this link has not been established in the ESRD population.

Comparisons: The amount of muscle fatigue during intermittent submaximal quadriceps exercise between dialysis patients and controls will be compared. In addition, the degree of exercise-induced increase in markers of oxidative stress in muscle and in plasma will be compared between dialysis patients and controls and between dialysis patients who have received N-acetylcysteine for 6 days and those who have received placebo capsules.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* undergoing hemodialysis for 3 months or more or healthy control without kidney disease

Exclusion Criteria:

* inability to give informed consent
* diagnosis of diabetes mellitus
* musculoskeletal contraindication to exercise
* infection requiring intravenous antibiotics within 2 months
* hospitalization within 2 months
* ingestion of antioxidant supplements within one month
* requirement for systemic anticoagulation
* estimated GFR <60 ml/min/1.73 m2 for healthy controls

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
change in quadriceps muscle endurance during intermittent submaximal contractions | 6 days
change in exercise-induced markers of oxidative stress | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten L Johansen, MD, Principal Investigator — University of California, San Francisco, San Francisco VA Medical Center
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553